CLINICAL TRIAL: NCT04238481
Title: A Phase 2 Randomized Open-label, Dose-ranging Study for Ureter Visualization Using ASP5354 in Subjects Undergoing Laparoscopic/Minimally Invasive Colorectal Surgery
Brief Title: A Study for Ureter Visualization, Using ASP5354 in Subjects Undergoing Laparoscopic/Minimally Invasive Colorectal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5354-CL-0201
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2023-08

CONDITIONS: Laparoscopic/Minimally Invasive Colorectal Surgery
Keywords: ASP5354; ureter visualization; imaging agent; near infrared fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pudexacianinium chloride - Dose Level A (Experimental): Participants received single dose of pudexacianinium chloride at dose level A by intravenous (IV) bolus infusion on day 1 once the surgical area of interest is in view.
  Interventions: Drug: Pudexacianinium chloride
- Pudexacianinium chloride - Dose Level B (Experimental): Participants received single dose of pudexacianinium chloride at dose level B by IV bolus infusion on day 1 once the surgical area of interest is in view.
  Interventions: Drug: Pudexacianinium chloride
- Pudexacianinium chloride - Dose Level C (Experimental): Participants received single dose of pudexacianinium chloride at dose level C by IV bolus infusion on day 1 once the surgical area of interest is in view.
  Interventions: Drug: Pudexacianinium chloride
- Pudexacianinium chloride - Dose Level B - Dose Expansion (Experimental): Participants who were enrolled in the dose expansion group received single dose of pudexacianinium chloride at dose level B by IV bolus infusion on day 1 once the surgical area of interest is in view.
  Interventions: Drug: Pudexacianinium chloride

INTERVENTIONS:
Drug: Pudexacianinium chloride — Intravenous
  Other Names: ASP5354

SUMMARY:
The primary purpose of this study was to determine the optimal dose of ASP5354 for ureter visualization in participants undergoing laparoscopic/minimally invasive colorectal surgery This study also investigated the safety, tolerability and the pharmacokinetics of ASP5354 in participants undergoing laparoscopic/minimally invasive colorectal surgery.

DETAILED DESCRIPTION:
Participants were randomly assigned at each dose level (dose A, B, C). During a standard minimally invasive surgery, visualization of the surgical field was assessed following the placement of the near infrared fluorescence (NIR F) imaging system proximal to the ureter of interest and then ASP5354 was administered.

Based on Visualization Review Committee (VRC) review of the initial 3 dose levels, if none of the doses selected had visualization, then additional two dose levels (dose D and E) was planned to be added; if 1 dose selected has visualization, then the dose level D was planned to be added. The dose level F was planned to be added if only the dose E level has visualization.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled to undergo laparoscopic/minimally invasive colorectal surgery.
* Subject will need visualization of the ureter(s).
* Female subject is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 30 days after final study treatment administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period.
* Female subject must not donate ova starting at first dose of investigational product (IP) and throughout the study period and for 30 days after final study treatment administration.
* Male subject with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 30 days after final study treatment administration.
* Male subject must not donate sperm during the treatment period and for 30 days after final study treatment administration.
* Male subject with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 30 days after final study treatment administration.
* Subject agrees not to participate in another interventional study while participating in the present study.
* Subjects enrolled after optimal dose determination:

Subject has any of the following values at screening:

* Body mass index > 25
* Estimated glomerular filtration rate (eGFR) ≥ 15 mL/min/1.73 m^2 and < 60. Subjects with an eGFR ≥ 60 mL/min/1.73 m^2 may be considered after discussion with the medical monitor.

Exclusion Criteria:

* Subject is anticipated to require ureteral stenting during surgery.
* Subject has a history of known retroperitoneal fibrosis.
* Subject has an active urinary tract infection.
* Subject has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subject has any condition that makes the subject unsuitable for study participation.
* Subject has a known or suspected hypersensitivity to ASP5354, indocyanine green (ICG) or any components of the formulation used.
* Subject has had previous exposure to ASP5354.
* Subject has moderate to severe cardiac disease that limits daily functioning (New York Heart Association Class III-IV) or other medical conditions that the investigator feels would impact safety or study compliance.
* Subject has a mean resting heart rate ≤ 45 bpm or ≥ 115 bpm, mean systolic blood pressure (SBP) ≥ 160 mmHg or mean diastolic blood pressure (DBP) ≥ 100 mmHg on day -1. If the mean blood pressure exceeds the limits above, repeat readings can be taken. Subject who has adequately controlled blood pressure is eligible.
* Subject has a mean corrected QT interval (Triplicate electrocardiogram [ECG]) using Fridericia's formula (QTcF) > 430 msec (for male subjects) and > 450 msec (for female subjects) on day -1. If the mean QTcF exceeds the limits above, the mean of 1 additional triplicate ECG may be taken.
* Subject has any of the following screening laboratory values:

  * Hemoglobin ≤ 9 g/dL
  * Absolute neutrophil count ≤ 1500/µL
  * Platelet count ≤ 100000/µL
  * eGFR < 60 mL/min/1.73 m^2 (Not applicable to subjects enrolled after optimal dose determination.)
  * Serum bilirubin ≥ 2 × upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) or serum glutamic oxaloacetic transaminase ≥ 2.5 × ULN
  * Alanine aminotransferase (ALT) or serum glutamic pyruvic transaminase ≥ 2.5 × ULN
* Subject has taken ICG or other near-infrared fluorescence (NIR)-F imaging agents within 48 hours prior to study treatment administration.
* Subject has taken diuretics or inhibitors of renal transporters defined by Food and Drug Administration (FDA) within 48 hours prior to study treatment administration.
* Subject has used any illicit drugs, unless legally prescribed and is not being abused (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) within 1 month prior to day -1.
* Subject has a history of alcohol abuse. Subject should not have consumed any alcohol within 48 hours of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Inc
Locations (2):
- United States (2):
  - Center for Colon and Rectal Surgery; AdventHealth Medical Group, Orlando, Florida
  - Ochsner Medical Center, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Albert M, Delgado-Herrera L, Paruch J, Gerritsen-van Schieveen P, Kishimoto T, Takusagawa S, Cai N, Fengler J, Raizer J. Pudexacianinium (ASP5354) chloride for ureter visualization in participants undergoing laparoscopic, minimally invasive colorectal surgery. Surg Endosc. 2023 Sep;37(9):7336-7347. doi: 10.1007/s00464-023-10193-9. Epub 2023 Jul 20. PMID 37474823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants undergoing laparoscopic/minimally invasive colorectal surgery in which the need for anatomical visualization of the ureter was anticipated were enrolled into this study.
Pre-assignment Details: Eligible participants who met inclusion criteria and none of the exclusion criteria were enrolled. A total of 13 participants were randomized, of which 12 participants received study drug.
Groups:
- Pudexacianinium Chloride - Dose Level A: Participants received single dose of pudexacianinium chloride at dose level A by IV bolus infusion on day 1 once the surgical area of interest is in view.
Period: Overall Study
Arm/Group | Pudexacianinium Chloride - Dose Level A | Pudexacianinium Chloride - Dose Level B | Pudexacianinium Chloride - Dose Level C | Pudexacianinium Chloride - Dose Level B - Dose Expansion
Started | 3 | 4 | 3 | 3
Treated | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 1 | 0 | 0
Not completed — Miscellaneous | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all randomized participants who received pudexacianinium chloride and had at least 1 assessment of ureter visualization during surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pudexacianinium Chloride - Dose Level A | Pudexacianinium Chloride - Dose Level B | Pudexacianinium Chloride - Dose Level C | Pudexacianinium Chloride - Dose Level B - Dose Expansion | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (2.5) | 56.7 (11.6) | 38.3 (12.4) | 57.3 (5.7) | 51.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 3 | 10
  Male | 0 | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 0 | 4
  Not Hispanic or Latino | 2 | 1 | 2 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 2 | 3 | 3 | 2 | 10
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Anatomical Visualization of the Index Ureter(s)
Description: The anatomical visualization of the index ureter(s) was assessed by the investigator intraoperatively using a binary "Yes or No" question on the ability to visualize the ureter and was assessed as successful, if both 30 minutes after pudexacianinium chloride dosing and at end of surgery the visualization was assessed as positive (Yes)/successful. For imputation of missing values at 30 minutes after pudexacianinium chloride administration, the nearest time points before and after the 30 minutes was considered. If both time points (before and after 30 minutes) were successful, 30 minutes anatomical visualization was imputed as successful. If both time points were not successful, then 30 minutes anatomical visualization was imputed as not successful, and all other cases were not imputed.
Time Frame: 30 minutes postdose through end of surgery (on day 1)
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pudexacianinium Chloride - Dose Level A | Pudexacianinium Chloride - Dose Level B | Pudexacianinium Chloride - Dose Level C | Pudexacianinium Chloride - Dose Level B - Dose Expansion
Number analyzed (Participants) | 3 | 3 | 3 | 3
percentage of participants | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 66.7 [9.4 to 99.2]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered an investigational product (IP), and which did not necessarily have a causal relationship with the treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP whether or not considered related to the IP. A TEAE was defined as an AE observed after administration of the IP and up to the follow-up period. An AE was considered "serious" if the event: results in death;is life-threatening; results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions;results in congenital anomaly, or birth defect;requires inpatient hospitalization (except for planned procedures as allowed per study) or leads to prolongation of hospitalization; Other medically important events.
Time Frame: From first dose of study drug until follow-up period (day 10)
Population: The safety analysis set (SAF) consisted of all randomized participants who received pudexacianinium chloride.
Measure: Number; unit: participants
Arm/Group | Pudexacianinium Chloride - Dose Level A | Pudexacianinium Chloride - Dose Level B | Pudexacianinium Chloride - Dose Level C | Pudexacianinium Chloride - Dose Level B - Dose Expansion
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 2 | 2 | 1 | 1

3. Secondary Outcome: Plasma Concentration of Pudexacianinium Chloride
Description: Plasma concentration of pudexacianinium chloride was reported from the blood samples collected. Concentrations below the lower limit of quantification (1 nanogram per milliliter [ng/mL]) are set to zero.
Time Frame: Predose, 10, 30, 60, 90, 120 minutes, end of surgery, 180 mins post dose
Population: The pharmacokinetic analysis set (PKAS) consisted of all randomized participants who received pudexacianinium chloride and had at least 1 plasma or urine concentration data available with the time of dosing and sampling. Participants with available data at specified time point were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pudexacianinium Chloride - Dose Level A | Pudexacianinium Chloride - Dose Level B | Pudexacianinium Chloride - Dose Level C | Pudexacianinium Chloride - Dose Level B - Dose Expansion
Number analyzed (Participants) | 3 | 3 | 3 | 3
ng/mL
  Predose | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  10 Minutes | 48.9 (20.6) | 196 (161) | 322 (177) | 272 (278)
  30 Minutes: number analyzed (Participants) | 3 | 3 | 3 | 2
  30 Minutes | 22.5 (3.30) | 58.0 (5.74) | 146 (46.1) | 81.1 (16.2)
  60 Minutes: number analyzed (Participants) | 1 | 2 | 1 | 0
  60 Minutes | 15.3 | 38.2 (7.35) | 106 |
  90 Minutes: number analyzed (Participants) | 1 | 1 | 0 | 0
  90 Minutes | 12.7 | 34.4 |  |
  120 Minutes: number analyzed (Participants) | 1 | 0 | 0 | 0
  120 Minutes | 8.37 |  |  |
  End of Surgery: number analyzed (Participants) | 3 | 3 | 2 | 3
  End of Surgery | 14.0 (5.98) | 28.0 (1.64) | 47.3 (29.8) | 51.0 (14.7)
  180 Minutes: number analyzed (Participants) | 0 | 1 | 0 | 1
  180 Minutes |  | 18.0 |  | 41.5

4. Secondary Outcome: Urine Concentration of Pudexacianinium Chloride
Description: Urine concentration of pudexacianinium chloride was reported from the urine samples collected. Concentrations below the lower limit of quantification (20 ng/mL) are set to zero.
Time Frame: Predose, 10, 30, 60, 90 minutes, end of surgery, 180 mins post dose
Population: PKAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pudexacianinium Chloride - Dose Level A | Pudexacianinium Chloride - Dose Level B | Pudexacianinium Chloride - Dose Level C | Pudexacianinium Chloride - Dose Level B - Dose Expansion
Number analyzed (Participants) | 3 | 3 | 2 | 3
ng/mL
  Predose | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  10 Minutes: number analyzed (Participants) | 1 | 2 | 0 | 0
  10 Minutes | 0 | 695 (983) |  |
  30 Minutes: number analyzed (Participants) | 0 | 2 | 0 | 0
  30 Minutes |  | 10800 (8620) |  |
  60 Minutes: number analyzed (Participants) | 0 | 2 | 0 | 0
  60 Minutes |  | 12000 (7420) |  |
  90 Minutes: number analyzed (Participants) | 0 | 1 | 0 | 0
  90 Minutes |  | 6800 |  |
  End of Surgery: number analyzed (Participants) | 2 | 2 | 2 | 0
  End of Surgery | 1960 (955) | 4840 (3650) | 33800 (636) |
  180 Minutes: number analyzed (Participants) | 0 | 1 | 0 | 0
  180 Minutes |  | 953 |  |

5. Secondary Outcome: Amount of Pudexacianinium Chloride Excreted in Urine (Ae) During Surgery
Description: Amount of pudexacianinium chloride excreted in urine during surgery was reported.
Time Frame: During surgery (on day 1)
Population: PKAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Pudexacianinium Chloride - Dose Level A | Pudexacianinium Chloride - Dose Level B | Pudexacianinium Chloride - Dose Level C | Pudexacianinium Chloride - Dose Level B - Dose Expansion
Number analyzed (Participants) | 3 | 2 | 3 | 1
milligrams (mg) | 0.0670 (0.0239) | 0.212 (0.0339) | 1.19 (0.371) | 0.0438

6. Secondary Outcome: Percentage of Pudexacianinium Chloride Dose Excreted Into Urine (Ae%) During Surgery
Description: Percentage of pudexacianinium chloride dose excreted into urine during surgery was reported.
Time Frame: During surgery (on day 1)
Population: PKAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: percentage of drug excreted
Arm/Group | Pudexacianinium Chloride - Dose Level A | Pudexacianinium Chloride - Dose Level B | Pudexacianinium Chloride - Dose Level C | Pudexacianinium Chloride - Dose Level B - Dose Expansion
Number analyzed (Participants) | 3 | 2 | 3 | 1
percentage of drug excreted | 22.3 (7.98) | 21.2 (3.39) | 39.5 (12.4) | 4.38

ADVERSE EVENTS:
Time Frame: From first dose of study drug until follow-up period (day 10)
Description: SAF Population
Groups:
- Pudexacianinium Chloride - Dose Level C: Participants received single dose pudexacianinium chloride at dose level C by IV bolus infusion on day 1 once the surgical area of interest is in view.
Arm/Group | Pudexacianinium Chloride - Dose Level A | Pudexacianinium Chloride - Dose Level B | Pudexacianinium Chloride - Dose Level C | Pudexacianinium Chloride - Dose Level B - Dose Expansion
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 1/3 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pudexacianinium Chloride - Dose Level A (N=3) | Pudexacianinium Chloride - Dose Level B (N=3) | Pudexacianinium Chloride - Dose Level C (N=3) | Pudexacianinium Chloride - Dose Level B - Dose Expansion (N=3)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pudexacianinium Chloride - Dose Level A (N=3) | Pudexacianinium Chloride - Dose Level B (N=3) | Pudexacianinium Chloride - Dose Level C (N=3) | Pudexacianinium Chloride - Dose Level B - Dose Expansion (N=3)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT04238481/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT04238481/SAP_001.pdf